CLINICAL TRIAL: NCT02260687
Title: Special Drug Use Investigation of EYLEA for Myopic Choroidal Neovascularization
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 17416; EY1414JP (Other: Company Internal)
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Choroidal Neovascularization
Keywords: Aflibercept; Anti-VEGF
MeSH Terms: conditions — Choroidal Neovascularization | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Decision of treatment is made by attending investigator according to the Japanese Package Insert
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Administration by intravitreal injection

SUMMARY:
The objectives of this study are to investigate the safety and effectiveness of EYLEA.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, multi center post-authorization safety study that includes patients with a diagnosis of myopic choroidal neovascularization. The investigator will have made the choice of treatment (EYLEA) as well as the decision to use EYLEA according the Japanese Package Insert prior to enrolling the patient in this study.

The observation period for each patient starts when therapy with EYLEA is initiated. The enrollment period is 2 years. Patients will be followed for a time period of 1 years or until it is no longer possible (e.g. lost to follow-up within the 1 year ). In total, 300 patients will be recruited.

For each patient, data are collected as defined in the electronic case report form (eCRF) at the initial visit, follow-up visits and final visit, either by routine clinical visits (as per investigators routine practice) .

ELIGIBILITY:
Inclusion Criteria:

* Patients who start EYLEA treatment for mCNV(myopic choroidal neovascularization).

Exclusion Criteria:

* Patients who have already received EYLEA treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female and male patients with mCNV(myopic choroidal neovascularization) diagnosis will be enrolled after the investigators have taken the decision for the treatment with EYLEA. Those patients who have had EYLEA prescribed previously will not be included in this study. Physicians should consult the full prescribing information for EYLEA before enrolling patients and be familiarized with the safety information in the product package label.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Number of episodes of Adverse drug reaction (ADR's) | Up to 12 months
Number of episodes of Infections | Up to 12 months
Number of episodes of Serious Adverse Events(SAE's) | Up to 12 months
Number of episodes of Ocular Adverse events | Up to 12 months

SECONDARY OUTCOMES:
Mean changes in visual acuity | Baseline up to 12 months
Mean changes in retina thickness | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Japan

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/